CLINICAL TRIAL: NCT06389292
Title: A Global, Multicenter, Randomized, Double-blind, Phase 3 Pivotal Registrational Clinical Study of APG-2575 (Lisaftoclax) Combined With Azacitidine in Elderly Patients With Newly Diagnosed Acute Myeloid Leukemia (GLORA-3)
Brief Title: A Pivotal Study of APG-2575 (Lisaftoclax) Combined With Azacitidine in the Treatment of Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APG2575AG301
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: APG -2575; Lisaftoclax
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Lisaftoclax; Azacitidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APG-2575 (Lisaftoclax) combined with Azacitidine (Experimental)
  Interventions: Drug: APG-2575(Lisaftoclax ); Drug: Azacitidine Injection
- Placebo combined with Azacitidine (Active Comparator)
  Interventions: Other: Placebo; Drug: Azacitidine Injection

INTERVENTIONS:
Drug: APG-2575(Lisaftoclax ) — QD, oral administration, every 28 days for a dosing cycle.
  Arms: APG-2575 (Lisaftoclax) combined with Azacitidine
Other: Placebo — QD, oral administration, every 28 days for a dosing cycle.
  Arms: Placebo combined with Azacitidine
Drug: Azacitidine Injection — QD, subcutaneous or intravenous injection, D1-7 in 28-day cycle.

SUMMARY:
A global, multicenter, randomized, double-blind, placebo-controlled, phase III pivotal registration study, to evaluate the efficacy of APG-2575 (Lisaftoclax) combined with azacitidine (AZA) versus placebo combined with azacitidine in newly diagnosed acute myeloid leukemia who are not eligible for standard induction chemotherapy.

DETAILED DESCRIPTION:
The newly diagnosed acute myeloid leukemia, who are not eligible for standard induction chemotherapy, will be randomized to the investigational group 'Lisaftoclax (APG-2575) + AZA' or the control group 'placebo+ AZA'.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have newly diagnosed AML that meets the criteria for acute myeloid leukemia (AML) and ineligible for standard chemotherapy.
2. Life expectancy of ≥3 months.
3. Be able to accept oral administration.
4. Patients aged ≥70 years with ECOG score of 0-2, or those aged≥18 years and <70 years with ECOG score of 0-3.
5. Adequate kidney function.
6. White blood cell ≤ 30×10^9/L.
7. Adequate liver function.
8. Men, women with childbearing potential, and their partners voluntarily use contraception that researchers consider effective.
9. Be able to understand and voluntarily sign written informed consent.
10. Patients must be willing and able to complete study procedures and follow-up examinations.

Exclusion Criteria:

1. The patient was diagnosed with acute promyelocytic leukemia or AML BCR-ABL1 positive.
2. Active leukemic infiltration of the central nervous system.
3. Active infection that is uncontrolled and requires systemic treatment.
4. Use of strong inducers of CYP3A4 within 7 days prior to the first dose of the investigational drug, and/or use of moderate to strong inhibitors of CYP3A4 within 7 days or 3-5 half-lives (whichever is longer) prior to the first dose of the investigational drug.
5. Previous treatment for hematologic disorders.
6. Patients who has a cardiovascular disability status of New York Heart Association Class > 2.
7. Patients have malabsorption syndrome or other conditions that cannot be administered through the gastrointestinal tract or affect drug absorption.
8. Patients had a history of other malignancies prior to study initiation.
9. Any other circumstances or conditions, at the discretion of the investigator, make the patient unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2028-05-25 (Estimated); Study Completion 2029-03-26 (Estimated)

PRIMARY OUTCOMES:
Overall Survival（OS） | Up to 5 years
  The primary endpoint was overall survival (OS), defined as the time from the date of randomization to the date of death of any cause.

SECONDARY OUTCOMES:
Percentage of Participants with Objective Response Rate (ORR) | Up to 5 years
  ORR is defined as the proportion of patients who have achieved CR, CRi, CRh, MLFS or PR.
Safety evaluation based on the adverse event concurrence | Up to 5 years
  Number of treatment emergent adverse events (TEAEs) and treatment related adverse events (TRAEs) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, M.D., Principal Investigator — Hematology Hospital of the Chinese Academy of Medical Sciences; Jie Jin, M.D., Principal Investigator — Zhejiang University
Locations (6):
- China (2):
  - Hematology Hospital of the Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Russia (4):
  - Moscow Multidisciplinary Clinical Center "Kommunarka", Moscow
  - Botkin Moscow Multidisciplinary Research and Clinical Center, Moscow
  - Russian Research Institute of Hematology and Transfusiology of the Federal Medical and Biological Agency, Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg